CLINICAL TRIAL: NCT05615753
Title: Feasibility of Implementing Acupuncture Into a Federally Qualified Health Center to Alleviate Multiple Symptoms Among Breast Cancer Survivors
Brief Title: Feasibility of Implementing Acupuncture Into Federally Qualified Health Center Among Breast Cancer Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Hongjin Li, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-0353
Record Dates: First submitted 2022-10-25; First posted 2022-11-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Experimental): Participants will receive 2 acupuncture treatments each week for 5 weeks, for a total of 10 treatments. Each acupuncture treatment will take 30 minutes.
  Interventions: Behavioral: Acupuncture
- Usual care group (No Intervention): Participants will continue to receive their usual care.

INTERVENTIONS:
Behavioral: Acupuncture — All participants will receive a semi-standardized acupuncture protocol with additional points for patient's particular pain location,
  Arms: Acupuncture group

SUMMARY:
The purpose of this study is to test the feasibility of implementing acupuncture intervention in federally qualified health centers oncology clinics for breast cancer survivors.

DETAILED DESCRIPTION:
This study has the following specific aims:

Aim 1: Test the feasibility and acceptability of implementing a 5-week acupuncture intervention within federally qualified health center oncology clinic to manage multiple symptoms (pain, hot flashes, fatigue, sleep disturbance, depression, anxiety) among breast cancer survivors receiving endocrine therapy.

Aim 2: Use a mixed methods approach to identify barriers and facilitators associated with implementing acupuncture in federally qualified health center oncology clinic.

ELIGIBILITY:
Inclusion Criteria:

* women with histologically confirmed stage 0, I, II, or III breast cancer
* > 18 years of old
* who have completed their primary cancer treatment (e.g., surgery, radiotherapy, chemotherapy) in the past 1 month and currently taking endocrine therapy
* are able to read and speak English
* with self-reported pain, fatigue, sleep disturbance, depression, hot flashes and/or anxiety in the last month and their average severity rating ≥ 3 (0-10 numeric rating scale) for at least 3 of the 6 symptoms, and experience at least 2 physical symptoms (pain, fatigue, sleep disturbance).

Exclusion Criteria:

* Metastatic breast cancer (stage IV)
* have a bleeding disorder (e.g. hemophilia, Von Willebrand's disease, thrombocytopenia)
* failure to comply with weekly visits to the acupuncture clinic during the interventional phase of the study
* Psychiatric or medical disorders which would affect study assessments, such as, dementia, Alzheimer's disease, a history of any neurological condition, traumatic brain injury, stroke, and the use of psychotropic medication
* Breastfeeding, pregnant or are planning get pregnant during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Acceptability for Treating Multiple Symptoms with Acupuncture | At week 6 after finishing the 10th acupuncture treatment
  Protocol Acceptability Scale is a 9-item instrument with scores ranging from 0 to 18 used to measure acceptability of the study processes and protocols. Items are measured on a 0 to 2 scale, where 0 means "did not like the study/did not like acupuncture/did not enjoy participating", and 2 means "liked the study/liked acupuncture/enjoyed participating". The protocol was deemed to have high acceptability if 80% of participants scored ≥ 80% of possible points on the acceptability scale. The investigators calculated the mean score for each of the 9 questions, divided the total score for the 9 questions by the maximum possible points for the measure, and converted the total mean scores to percentage of participants who liked the study/liked acupuncture/enjoyed participating.
The numbers of study participants being recruited and retained (Feasibility) | : from the activation of the study to the completion of the recruitment, week 12
  The numbers of study participants being recruited and retained during the study period will be documented as planned
Identify barriers and facilitators associated with implementing acupuncture in federally qualified health center oncology clinics. | Through study completion, an average of 1 year
  Specific questions will be asked during a face-to-face interview to identify factors favoring or barriers to implementing acupuncture into federally qualified health center oncology clinics among breast cancer survivors and providers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No